CLINICAL TRIAL: NCT05131022
Title: A Phase 1, Dose Escalation, and Cohort Expansion Study Evaluating NX-5948, a Bruton's Tyrosine Kinase (BTK) Degrader, in Adults With Relapsed/Refractory B-cell Malignancies
Brief Title: A Study of NX-5948 in Adults With Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NX-5948-301; 2023-510541-25-00 (EU CTIS Number); 2021-003125-29 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Diffuse Large B Cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); Waldenstrom Macroglobulinemia (WM); Primary Central Nervous System Lymphoma (PCNSL); Secondary Central Nervous System Lymphoma (SCNSL)
Keywords: BTK Degrader; BTK Inhibitor; B-Cell Malignancy; Lymphoma; C481; C481S; Bruton's Tyrosine Kinase; NX-5948; Targeted Protein Degradation; Chimeric Targeting Molecule (CTM)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (19):
- Phase 1a Dose Escalation (Experimental): Multiple dose levels of NX-5948 to be evaluated; determination of Maximum Tolerated Dose/Phase 1b recommended dose(s)
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 1 in CLL or SLL with prior BTKi and BCL2i (Experimental): CLL or SLL with prior exposure to both a Bruton's tyrosine kinase inhibitor (BTKi) and BCL-2 inhibitor, unless previously deemed ineligible for a BCL-2i. Patients enrolled in CLL/SLL arm will be randomized to one of two dose levels.
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 2 in CLL/SLL with non-C481S BTK mutations (Experimental): Prior exposure to both BTKi and BCL-2i (unless deemed ineligible for BCL-2i by Investigator at the time of study enrollment) and documented BTK mutation other than C481S within 6 months prior to study entry
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 3 in CLL/SLL with prior non-covalent BTKi (Experimental): CLL/SLL with prior exposure to ncBTKi and are BCL-2i naïve.
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 4 in CLL/SLL with TP53 or 17p deletion, 2L, prior BTKi (Experimental): Patients with documented TP53 mutation or 17p deletion and 1 prior line of therapy that included a BTKi and are BCL-2i naïve.
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 5 in CLL/SLL with 2L+, prior BTKi (Experimental): Patients with at least 1 prior line of therapy that included a BTKi and are BCL-2i naïve.
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 6 in MCL (Experimental): Non-blastoid MCL with prior exposure to a BTKi and an anti-CD20 monoclonal antibody (mAb)-based chemoimmunotherapy regimen
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 7 in MZL (Experimental): MZL (EMZL, MALT, NMZL, SMZL) with prior exposure to an anti-CD20 mAb-based chemo-immunotherapy regimen and an additional line of therapy
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 8 in WM (3L+) (Experimental): WM with prior exposure to a BTKi and at least an additional line of therapy
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 9 in WM (2L) (Experimental): WM following upfront therapy with a BTKi
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 10 in DLBCL (Experimental): DLBCL which transformed from indolent lymphoma or Richters transformation with prior exposure to an anthracycline (unless previously deemed ineligible to receive), an anti-CD20 mAb-based chemoimmunotherapy regimen, and an additional line of therapy
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 11 in FL (Experimental): FL (grade 1-3a) with prior exposure to an anti-CD20 mAb-based chemoimmunotherapy regimen and an additional line of therapy
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 12 in PCNSL/SCNSL (Experimental): PCNSL following at least 1 prior line of therapy that included a BTKi (2L+) or following 2 or more prior lines of therapy (3L+), or SCNSL patients meeting criteria for a non-CLL/SLL cohort enrolling that disease with secondary CNS involvement of lymphoma
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 13 in PCNSL (Experimental): PCNSL following upfront therapy and with no prior exposure to a BTKi (2L).
  Interventions: Drug: NX-5948
- Phase 1b Part 2 in CLL or SLL with prior BTKi and BCL-2i (Experimental): CLL or SLL with prior exposure to both a Bruton's tyrosine kinase inhibitor (BTKi) and BCL-2 inhibitor
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 14 in first-line WM (Experimental): Treatment-naïve WM deemed unfit for chemoimmunotherapy
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 15 in BTKi-naive CLL/SLL (Experimental): First-line (1L) or second-line+ (2L)+ CLL/SLL with no prior exposure to a BTKi
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 16 in CLL/SLL with secondary warm autoimmune hemolytic anemia (wAIHA) (Experimental): BTKi-exposed R/R CLL or SLL with secondary wAIHA
  Interventions: Drug: NX-5948
- Phase 1b Part 1 Cohort 17 in CLL/SLL with CNS involvement (Experimental): BTKi-exposed R/R CLL or SLL with CNS involvement
  Interventions: Drug: NX-5948

INTERVENTIONS:
Drug: NX-5948 — Oral NX-5948

SUMMARY:
This is a first-in-human Phase 1a/1b multicenter, open-label study designed to evaluate the safety and anti-cancer activity of NX-5948 in patients with advanced B-cell malignancies.

DETAILED DESCRIPTION:
Phase 1a is a dose escalation to evaluate the safety and tolerability of NX-5948 in adult patients with relapsed/refractory (R/R) B cell malignancies who have received at least 2 prior lines of therapy, or at least 1 prior line of therapy for Primary Central Nervous System Lymphoma (PCNSL), and for whom no other therapies are known to provide clinical benefit. Indications include: Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL), Diffuse Large B-cell Lymphoma (DLBCL), Mantle Cell Lymphoma (MCL), Waldenstrom Macroglobulinemia (WM), Marginal Zone Lymphoma (MZL), Follicular Lymphoma (FL), Primary Central Nervous System Lymphoma (PCNSL) or any of the above indications with disease in the central nervous system or Secondary Central Nervous System Lymphoma (SCNSL).

Phase 1b Part 1, called safety expansion, investigates the safety and anti-tumor activity of NX-5948 at the dose(s) selected in Phase 1a in up to 17 expansion cohorts of patients with histologically confirmed B-cell malignancy indications who have received specified prior therapies based on indication:

* CLL or SLL (patients may be randomized to one of two dose levels investigated for CLL/SLL until an optimal dose is selected)
* MCL
* MZL
* WM
* DLBCL
* FL
* PCNSL/SCNSL

Phase 1b Part 2, called cohort expansion, will further investigate the anti-tumor activity of NX-5948 at the dose(s) selected in Phase 1b par 1 in one additional expansion arm of CLL/SLL patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years
* Patients in Phase 1a (Dose Escalation) must have histologically confirmed R/R CLL, SLL, DLBCL (subgroups include Richter-transformed DLBCL, germinal center B-cell type, activated B-cell type, high-grade B-cell lymphoma with MYC and BCL-2 and/or BCL-6 rearrangements, high-grade B-cell lymphomas NOS), FL, MCL, MZL (subtypes include EMZL, MALT, NMZL, SMZL), WM, or PCNSL.
* Patients in Phase 1a must meet the following:

  o For non-PCNSL indications, received at least 2 prior lines of therapy and have no other available therapies known to provide clinical benefit. For PCNSL, received at least 1 prior line of therapy
* Patients in Phase 1b (Safety and Cohort Expansion) must have 1 of the following histologically documented B-cell malignancies, must meet criteria for systemic treatment, and must have received prior therapies and/or molecular features based on details described for each cohort: CLL or SLL, DLBCL, MCL, FL, MZL, WM, or PCNSL/SCNSL.
* Measurable disease per response criteria specific to the malignancy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (0-2 for patients with PCNSL and secondary CNS involvement).
* Adequate organ and bone marrow function

Key Exclusion Criteria:

* Known or suspected active prolymphocytic leukemia or Richter's transformation to Hodgkin's lymphoma prior to study enrollment
* Prior treatment for the indication under study for anti-cancer intent that includes:

  1. Radiotherapy within 2 weeks of planned start of study drug (excluding limited palliative radiation).
  2. Prior systemic chemotherapy within 2 weeks of planned start of study drug.
  3. Prior monoclonal antibody therapy within 4 weeks of planned start of study drug, except for patients enrolling in Cohort 16 (CLL with secondary wAIHA) where a 16-week washout period is required.
  4. Prior small molecule therapy within 2 weeks or 5 half-lives (whichever is shorter) of planned start of study drug.
  5. Autologous or allogeneic stem cell transplant within 100 days prior to planned start of study drug.
  6. Chimeric antigen receptor (CAR) T-cell therapy within 100 days prior to start of study drug (within 60 days prior to start of study drug for Phase 1b).
  7. Use of systemic corticosteroids outside of dosing limits described below and within 7 days prior to initiation of study treatment excepting those used as prophylaxis for radio diagnostic contrast. Patients with PCNSL/SCNSL: no greater than 40 mg/day prednisone, or equivalent. Patients with PCNSL/SCNSL using greater than 20 mg/day prednisone, or equivalent, must be clinically stable at that dose for 7 days. All other diagnoses: no greater than 20 mg/day prednisone or equivalent.
  8. Use of systemic immunosuppressive drugs other than systemic corticosteroids for any medical condition within 60 days prior to first dose of study drug
  9. Previously treated with a BTK degrader
* Active, uncontrolled autoimmune hemolytic anemia (except for patients enrolling in Cohort 16) or active, uncontrolled autoimmune thrombocytopenia.
* Patient has any of the following within 6 months of planned start of study drug:

  1. Myocardial infarction, unstable angina, unstable symptomatic ischemic heart disease, or placement of a coronary arterial stent
  2. Uncontrolled atrial fibrillation or other clinically significant arrhythmias, conduction abnormalities, or New York Heart Association (NYHA) class III or IV heart failure
  3. Thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), stroke, or intracranial hemorrhage
  4. Any other significant cardiac condition (e.g., pericardial effusion, restrictive cardiomyopathy, severe untreated valvular stenosis, severe congenital heart disease, or persistent uncontrolled hypertension defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg despite optimal medical management)
* Bleeding diathesis, or other known risk for acute blood loss.
* History of Grade ≥ 2 hemorrhage within 28 days of planned start of study drug.
* Active known concurrent malignancy or malignancy other than the one under study within the past 3 years. (Exceptions include, but are not limited to, patients with more recent history of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast may enroll if they have undergone curative therapy and have no evidence of disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with protocol specified dose-limiting toxicities | Up to 24 months
  Phase 1a
To establish the maximum tolerated dose and/or recommended Phase 1b dose(s) | Up to 24 months
  Phase 1a
To evaluate the anti-tumor activity of NX-5948 in the dose levels selected for Phase 1b safety expansion based on overall response rate (ORR) as assessed by Investigator | Up to 3 years
  Phase 1b Part 1
Number of participants with treatment-emergent adverse events (TEAEs); Grade 3, 4, 5 TEAEs, serious adverse events (SAEs), TEAEs leading to study drug discontinuation, deaths due to TEAEs, and all deaths | Up to 6 years
  Phase 1a / Phase 1b Part 1
To further evaluate the anti-tumor activity of NX-5948 in patients with CLL/SLL at the dose identified in Phase 1b Part 1 based on overall response rate (ORR) as assessed by Investigator | Up to 3 years
  Phase 1b Part 2

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of NX-5948: Maximum Serum Concentration | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2 - Sampling following the first dose, pre- and post-dose at selected cycles and at the end of treatment
Pharmacodynamic (PD) profile of NX-5948: Changes from baseline of BTK levels in B-cells | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2 - Sampling at screening, following the first dose, pre and post-dose at selected cycles and at the end of treatment
Complete response (CR) rate / CR with incomplete marrow recovery as assessed by the Investigator | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2
Duration of response (DOR) as assessed by the Investigator | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2
Progression-free survival (PFS) as assessed by the Investigator | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2
Time to next therapy | Up to 6 years
  Phase 1a / Phase 1b Part 1 and Part 2
Number of participants with treatment-emergent adverse events (TEAEs); Grade 3, 4, 5 TEAEs, serious adverse events (SAEs), TEAEs leading to study drug discontinuation, deaths due to TEAEs, and all deaths | Up to 3 years
  Phase 1b Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nurix Therapeutics, Inc.
Locations (62):
- United States (18):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - National Institute of Health, Bethesda, Maryland
  - Cayuga Medical Center, Ithaca, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (7):
  - CHU Angers, Angers
  - Hôpital Avicenne, Bobigny
  - CHU de Nantes, Nantes
  - CHU Bordeaux, Pessac
  - CHU de Poitiers, Poitiers
  - Institut Curie-Site Saint-Cloud, Saint-Cloud
  - CHRU de Nancy, Vandœuvre-lès-Nancy
- Italy (5):
  - IRCCS - AOU di Bologna, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - IRCCS Ospedale San Raffaele - Università Vita-Salute San Raffaele di Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
- Netherlands (4):
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Poland (7):
  - AidPort sp. Zo.o, Skórzewo, Greater Poland Voivodeship
  - Pratia MCM, Krakow, Lesser Poland Voivodeship
  - University Clinical Hostpital in Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - Pratia MTZ, Warsaw, Masovian Voivodeship
  - National Institute of Oncology Warszawa, Warsaw, Masovian Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
  - Medical University of Lublin, Lublin
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Cabuenes, Gijón
  - Hospital Ramón y Cajal, Madrid
  - Hospital Fundación Jimenez Díaz - START Madrid, Madrid
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital - Universitatsklinik Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- United Kingdom (10):
  - The Beatson WOS Cancer Center, Glasgow, Scotland
  - St. James Hospital, Leeds
  - Clatterbridge Cancer Center NHS Foundation Trust, Liverpool
  - St. Bartholomew's Hospital, Barts NHS Trust, London
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang D, Harris HM, Chen J, Judy J, James G, Kelly A, McIntosh J, Tenn-McClellan A, Ambing E, Tan YS, Lu H, Gajewski S, Clifton MC, Yung S, Robbins DW, Pirooznia M, Skanland SS, Gaglione E, Mhibik M, Underbayev C, Ahn IE, Sun C, Herman SEM, Noviski M, Wiestner A. NRX-0492 degrades wild-type and C481 mutant BTK and demonstrates in vivo activity in CLL patient-derived xenografts. Blood. 2023 Mar 30;141(13):1584-1596. doi: 10.1182/blood.2022016934. PMID 36375120